CLINICAL TRIAL: NCT07349654
Title: Underdilated-stent Technique Improves Post-transjugular Intrahepatic Portosystemic Shunt Encephalopathy: a Randomized Controlled Trial
Brief Title: Underdilated-stent Technique Improves Post-TIPS Encephalopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: West China Hospital (Other); Qianjiang Hospital, Chongqing University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UDS-TIPS-01
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Liver Cirrhosis; Variceal Bleeding, Cirrhosis; Ascites Hepatic; Hepatic Encephalopathy (HE)
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- underdilation group (Experimental): Patients in this group will receive a underdilated strategy during TIPS procedure by using a 6mm balloon to dilate the puncture tract and subsequently implanted 8mm Viatorr stent.
  Interventions: Device: 6mm balloon dilation
- full-dilation group (Active Comparator): Patients in this group will receive a fully-dilated strategy during TIPS procedure by using a 8mm balloon to dilate the puncture tract and subsequently implanted 8mm Viatorr stent.
  Interventions: Device: 8mm balloon dilation

INTERVENTIONS:
Device: 6mm balloon dilation — A 6mm balloon was used to under-dilate the puncture puncture tract and subsequently implanted 8mm Viatorr stent during TIPS procedure.
  Arms: underdilation group
Device: 8mm balloon dilation — A standard 8mm balloon was used to fully dilate the puncture puncture tract and subsequently implanted 8mm Viatorr stent during TIPS procedure.
  Arms: full-dilation group

SUMMARY:
Transjugular intrahepatic portosystemic shunt (TIPS) is a critical therapeutic approach for managing esophagogastric variceal bleeding and refractory ascites in decompensated cirrhosis patients. To date, hepatic encephalopathy (HE) remains one of the most common complications following TIPS procedures, and prediction and prevention of post-TIPS HE have always been a hotspot in the field of hepatology. However, no reliable clinical studies have confirmed that any drug or intervention can effectively prevent the occurrence of HE episodes following TIPS, including lactulose and rifaximin.

Underdilated strategy (UDS) was reported as an development technique proposed in recent years for TIPS procedures, which involves using a small-diameter balloon to dilate the puncture tract and subsequently implanted standard-diameter covered stent (e.g., 8 mm). This allows the stent to maintain a smaller diameter shortly after release, thereby reducing the incidence of hepatic encephalopathy during the postoperative period. Over time, the stent gradually dilates to its normal diameter within months. This period coincides with the higher incidence risk of post-TIPS HE, most commonly occurring within 6 months, especially within the first 3 months after TIPS. Therefore, theoretically, UDS can reduce the occurrence of post-TIPS HE. In terms of clinical research, however, there were still no high quality studies reported the advantages of this technique. Current reported clinical studies were all non-randomized controlled trials or retrospective studies, with low-quality evidence and sometimes contradictory findings.

The aim of this prospective randomized controlled clinical study is to evaluate whether administration of underdilated technology during TIPS can improve postoperative hepatic encephalopathy, without compromising the therapeutic efficacy of portal hypertension complications.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis, defined by clinical manifestations, biochemical indicators, imaging examinations, or liver biopsy;
* History of esophagogastric variceal bleeding, or refractory/recurrent ascites;
* Intended to undergo TIPS treatment.

Exclusion Criteria:

* Non-cirrhotic portal hypertension;
* Previous treatments that may affect portal pressure, such as TIPS or surgical procedures;
* History of overt hepatic encephalopathy (West-Haven classification ≥2);
* Malignant tumors in advanced stages;
* Concomitant irreversible heart, liver, kidney, or respiratory failure;
* Unable or unwilling to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of overt hepatic encephalopathy | 12 months
  West-Haven grade no less than 2.

SECONDARY OUTCOMES:
remission of complications of portal hypertention | 12 months
  variceal rebleeding diagnosed on endoscopy, or worsened ascites diagnosed by ultrasound or CT/MRI.
liver function | 12 months
  Child-Pugh Classification
liver transplantation-free survival | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Qianjiang Central Hospital, Qianjiang, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yao W, Liu JC, Wu YJ, Yang CT, Ju SG, Wang YL, Wang CY, Huang SJ, Bai YW, Chen Y, Li TQ, Zhou C, Xiong B. Effect of underdilated transjugular intrahepatic portosystemic shunt on prognosis in patients with prior splenectomy: a propensity score-matched case-control study. Abdom Radiol (NY). 2022 Oct;47(10):3615-3627. doi: 10.1007/s00261-022-03600-7. Epub 2022 Jul 12. PMID 35821274
- [Result] Gaba RC, Parvinian A, Minocha J, Casadaban LC, Knuttinen MG, Ray CE Jr, Bui JT. Should transjugular intrahepatic portosystemic shunt stent grafts be underdilated? J Vasc Interv Radiol. 2015 Mar;26(3):382-7. doi: 10.1016/j.jvir.2014.08.012. PMID 25735521
- [Result] Trebicka J, Bastgen D, Byrtus J, Praktiknjo M, Terstiegen S, Meyer C, Thomas D, Fimmers R, Treitl M, Euringer W, Sauerbruch T, Rossle M. Smaller-Diameter Covered Transjugular Intrahepatic Portosystemic Shunt Stents Are Associated With Increased Survival. Clin Gastroenterol Hepatol. 2019 Dec;17(13):2793-2799.e1. doi: 10.1016/j.cgh.2019.03.042. Epub 2019 Mar 30. PMID 30940552
- [Result] Luo X, Wang X, Zhu Y, Xi X, Zhao Y, Yang J, Li X, Yang L. Clinical Efficacy of Transjugular Intrahepatic Portosystemic Shunt Created with Expanded Polytetrafluoroethylene-Covered Stent-Grafts: 8-mm Versus 10-mm. Cardiovasc Intervent Radiol. 2019 May;42(5):737-743. doi: 10.1007/s00270-019-02162-4. Epub 2019 Jan 14. PMID 30643936
- [Result] Lv Y, Chen H, Luo B, Bai W, Li K, Wang Z, Xia D, Guo W, Wang Q, Li X, Yuan J, Cai H, Xia J, Yin Z, Fan D, Han G. Concurrent large spontaneous portosystemic shunt embolization for the prevention of overt hepatic encephalopathy after TIPS: A randomized controlled trial. Hepatology. 2022 Sep;76(3):676-688. doi: 10.1002/hep.32453. Epub 2022 Apr 15. PMID 35266571
- [Result] Yang M, Qiu Y, Wang W. Concurrent spontaneous portosystemic shunt embolization for the prevention of overt hepatic encephalopathy after TIPS: A systematic review and meta-analysis. Dig Liver Dis. 2024 Jun;56(6):978-985. doi: 10.1016/j.dld.2023.10.013. Epub 2023 Nov 3. PMID 37926635
- [Result] Bureau C, Thabut D, Jezequel C, Archambeaud I, D'Alteroche L, Dharancy S, Borentain P, Oberti F, Plessier A, De Ledinghen V, Ganne-Carrie N, Carbonell N, Rousseau V, Sommet A, Peron JM, Vinel JP. The Use of Rifaximin in the Prevention of Overt Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt : A Randomized Controlled Trial. Ann Intern Med. 2021 May;174(5):633-640. doi: 10.7326/M20-0202. Epub 2021 Feb 2. PMID 33524293
- [Result] Vilstrup H, Amodio P, Bajaj J, Cordoba J, Ferenci P, Mullen KD, Weissenborn K, Wong P. Hepatic encephalopathy in chronic liver disease: 2014 Practice Guideline by the American Association for the Study of Liver Diseases and the European Association for the Study of the Liver. Hepatology. 2014 Aug;60(2):715-35. doi: 10.1002/hep.27210. Epub 2014 Jul 8. No abstract available. PMID 25042402
- [Result] Riggio O, Nardelli S, Moscucci F, Pasquale C, Ridola L, Merli M. Hepatic encephalopathy after transjugular intrahepatic portosystemic shunt. Clin Liver Dis. 2012 Feb;16(1):133-46. doi: 10.1016/j.cld.2011.12.008. Epub 2012 Jan 4. PMID 22321469
- [Result] Riggio O, Ridola L, Lucidi C, Angeloni S. Emerging issues in the use of transjugular intrahepatic portosystemic shunt (TIPS) for management of portal hypertension: time to update the guidelines? Dig Liver Dis. 2010 Jul;42(7):462-7. doi: 10.1016/j.dld.2009.11.007. Epub 2009 Dec 29. PMID 20036625
- [Result] Yang Y, Liang X, Yang S, He X, Huang M, Shi W, Luo J, Duan C, Feng X, Fu S, Lu L. Preoperative prediction of overt hepatic encephalopathy caused by transjugular intrahepatic portosystemic shunt. Eur J Radiol. 2022 Sep;154:110384. doi: 10.1016/j.ejrad.2022.110384. Epub 2022 May 28. PMID 35667296
- [Result] Kabelitz MA, Sandmann L, Praktiknjo M, Mauz JB, Auer TA, Bruns T, Chang J, Engelmann C, Fehrenbach U, Hinrichs J, Jansen C, Kloeckner R, Kluwe J, Kohler M, Meyer C, Piecha F, Pollmanns MR, Ripoll C, Schultheiss M, Seifert LL, Stohr F, Sturm L, Trebicka J, Zipprich A, Labenz C, Bettinger D, Maasoumy B; German Cirrhosis Study Group. Early Occurrence of Hepatic Encephalopathy Following Transjugular Intrahepatic Portosystemic Shunt Insertion is Linked to Impaired Survival: A Multicenter Cohort Study. Clin Gastroenterol Hepatol. 2025 Nov;23(12):2214-2223.e27. doi: 10.1016/j.cgh.2025.01.024. Epub 2025 Mar 15. PMID 40097036
- [Result] Riggio O, Angeloni S, Salvatori FM, De Santis A, Cerini F, Farcomeni A, Attili AF, Merli M. Incidence, natural history, and risk factors of hepatic encephalopathy after transjugular intrahepatic portosystemic shunt with polytetrafluoroethylene-covered stent grafts. Am J Gastroenterol. 2008 Nov;103(11):2738-46. doi: 10.1111/j.1572-0241.2008.02102.x. Epub 2008 Sep 4. PMID 18775022
- [Result] Bureau C, Garcia-Pagan JC, Otal P, Pomier-Layrargues G, Chabbert V, Cortez C, Perreault P, Peron JM, Abraldes JG, Bouchard L, Bilbao JI, Bosch J, Rousseau H, Vinel JP. Improved clinical outcome using polytetrafluoroethylene-coated stents for TIPS: results of a randomized study. Gastroenterology. 2004 Feb;126(2):469-75. doi: 10.1053/j.gastro.2003.11.016. PMID 14762784
- [Result] Perarnau JM, Le Gouge A, Nicolas C, d'Alteroche L, Borentain P, Saliba F, Minello A, Anty R, Chagneau-Derrode C, Bernard PH, Abergel A, Ollivier-Hourmand I, Gournay J, Ayoub J, Gaborit C, Rusch E, Giraudeau B; STIC-TIPS group. Covered vs. uncovered stents for transjugular intrahepatic portosystemic shunt: a randomized controlled trial. J Hepatol. 2014 May;60(5):962-8. doi: 10.1016/j.jhep.2014.01.015. Epub 2014 Jan 27. PMID 24480619
- [Result] Gupta AC, Wang W, Shah C, Sands MJ, Bullen J, Remer EM, Bayona PM, Carey W, Kapoor B. Added Value of Covered Stents in Transjugular Intrahepatic Portosystemic Shunt: A Large Single-Center Experience. Cardiovasc Intervent Radiol. 2017 Nov;40(11):1723-1731. doi: 10.1007/s00270-017-1694-1. Epub 2017 May 16. PMID 28512687
- [Result] Wang Q, Lv Y, Bai M, Wang Z, Liu H, He C, Niu J, Guo W, Luo B, Yin Z, Bai W, Chen H, Wang E, Xia D, Li X, Yuan J, Han N, Cai H, Li T, Xie H, Xia J, Wang J, Zhang H, Wu K, Fan D, Han G. Eight millimetre covered TIPS does not compromise shunt function but reduces hepatic encephalopathy in preventing variceal rebleeding. J Hepatol. 2017 Sep;67(3):508-516. doi: 10.1016/j.jhep.2017.05.006. Epub 2017 May 12. PMID 28506905
- [Result] Dariushnia SR, Haskal ZJ, Midia M, Martin LG, Walker TG, Kalva SP, Clark TW, Ganguli S, Krishnamurthy V, Saiter CK, Nikolic B; Society of Interventional Radiology Standards of Practice Committee. Quality Improvement Guidelines for Transjugular Intrahepatic Portosystemic Shunts. J Vasc Interv Radiol. 2016 Jan;27(1):1-7. doi: 10.1016/j.jvir.2015.09.018. Epub 2015 Nov 21. No abstract available. PMID 26614596

DOCUMENTS (1):
  • Study Protocol (2024-09-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT07349654/Prot_000.pdf